CLINICAL TRIAL: NCT06010472
Title: An Exploratory Clinical Study of the Safety and Efficacy of Anti-CD19 Chimeric Antigen Receptor (CAR) Nature Killer Cells (KN5501) in the Treatment of Moderate to Severe Refractory Systemic Lupus Erythematosus (SLE)
Brief Title: An Exploratory Clinical Study of Anti-CD19 CAR NK Cells in the Treatment of Systemic Lupus Erythematosus
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: Rui Therapeutics Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHEC2023-174
Record Dates: First submitted 2023-08-07; First posted 2023-08-24 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2024-07

CONDITIONS: Systemic Lupus Erythematosus (SLE)
Keywords: Lupus Erythematosus, Systemic; Autoimmune disorders; Connective Tissue Diseases
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Autoimmune Diseases; Connective Tissue Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- anti-CD19 CAR NK cells (Experimental): To evaluate the safety and effectiveness of anti-CD19 CAR NK cells (KN5501) in patients with moderate to severe refractory SLE. All subjects will receive fludarabine/cyclophosphamide lymphodepletion followed by anti-CD19 CAR NK cells infusion.
  Interventions: Drug: anti-CD19 CAR NK cells (KN5501)

INTERVENTIONS:
Drug: anti-CD19 CAR NK cells (KN5501) — Patients will receive Fludarabine (25 mg/m2 per day) and Cyclophosphamide (300mg/m2 per day) on day -5, -4, and -3. Multiple doses of anti-CD19 CAR NK cells (KN5501) will infused in each group using the "3 + 3" dose-escalation strategy.

SUMMARY:
A single arm, open-label pilot study is designed to determine the safety and effectiveness of anti-cluster of differentiation antigen 19 (CD19) chimeric antigen receptor (CAR) natural killer (NK) cells (KN5501) in patients with moderate to severe refractory systemic lupus erythematosus (SLE). 36 patients are planned to be enrolled in the dose-escalation trial. The primary objective of the study was to evaluate the safety of allogeneic anti-CD19 CAR-NK cells (KN5501) for the treatment of patients with moderate to severe refractory active SLE. The secondary objective is to evaluate the efficacy of anti-CD19 CAR NK cells (KN5501) in patients with moderate to severe refractory SLE, including British Isles Lupus Assessment Group 2004 (BILAG-2004) index, Systemic Lupus Erythematosus Responder Index (SRI)-4 response rate, Lupus Low Disease Activity State (LLDAS) rate, and Definitions Of Remission In SLE (DORIS) remission rate.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 18 years old and ≤ 65 years old, male or female, subjects voluntarily participate in this clinical study and sign the Informed Consent Form (ICF)
2. Previous diagnosis of systemic lupus erythematosus (SLE) (according to the 1997 American Rheumatology Association criteria)
3. Females of childbearing potential must use effective contraception during study treatment and for 90 days after the last dose of study treatment. In addition, subjects must not donate eggs during the study and for at least 90 days after the last dose of study treatment
4. Subjects with Systemic Lupus Erythematosus Disease Activity Index (SLEDAI-2K) score ≥ 8 points prior to screening
5. Subject has ≥ 1 organ system with BILAG-2004 Class A mobility score or ≥ 2 organ systems with BILAG-2004 Class B mobility score prior to screening
6. Subjects meets one of the following:

   1. Antinuclear antibody (ANA) ≥ 1:80, determined by immunofluorescence method;
   2. Anti-dsDNA antibodies are higher than normal level;
   3. Anti-Smith antibodies are higher than normal level
7. Absolute number of neutrophils ≥ 1.0×10^9/L, hemoglobin ≥ 60g/L
8. Left ventricular ejection fraction (LVEF) ≥ 50%
9. Subjects have been treated with oral corticosteroids (OCS) in combination with an immunosuppressive or biologic agent for at least 6 months prior to enrollment

Exclusion Criteria:

1. Subjects with known severe allergic reactions, hypersensitivity, contraindication to any medications during the trial (cyclophosphamide, fludarabine, obinutuzumab), or subjects with a history of severe allergic reactions
2. Subjects with active infection receiving intravenous (IV) antibiotic treatment, or received intravenous (IV) antibiotic treatment within one week prior to anti-CD19 CAR NK Cells infusion
3. Subjects with acquired and congenital immunodeficiency diseases
4. Subjects with grade III or IV heart failure (NYHA classification)
5. History of epilepsy or other central nervous system (CNS) diseases
6. History of severe herpetic infection, such as herpetic encephalitis, ocular herpes, or diffuse herpes
7. History of other primary malignant tumors except:

   1. Cured non-melanoma skin cancer by surgical excision, for example basal cell carcinoma (BCC) ;
   2. Cured primary malignant tumors, such as cervical cancer, superficial bladder cancer, breast cancer
8. Signs of herpes or varicella-zoster virus infection (especially chickenpox, shingles) within 12 weeks prior to screening; History of any cardiac, endocrine, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, and renal disease or other major medical condition that would prevent the administration of anti-CD19 CAR NK Cells (KN5501), except for lupus (determined by the investigator)
9. Females who are pregnant, lactating, or planning a pregnancy within six months
10. Any active skin disease that may interfere with the study assessment of SLE, including but not limited to psoriasis, dermatomyositis, systemic sclerosis, non-LE cutaneous lupus manifestations (eg, cutaneous vascular disease, periungual telangiectasia, fingertip sclerosis, rheumatoid nodules, erythema multiforme, leg ulcers) or drug-induced lupus
11. Subjects who have received other clinical trial treatment within 3 months
12. Subjects who have received B cell-targeted drug therapy within 1 month before enrollment
13. Any abnormal laboratory test results judged by the investigator to be clinically significant and prevent the subject from participating in the study. Laboratory test values that are out of range and not of clinical significance will not be considered as exclusion criteria
14. Any situation judged by the investigators that may increase the risk of the subjects or interfere with the clinical trial outcome

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-08-20 (Actual); Primary Completion 2026-08-25 (Estimated); Study Completion 2027-08-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicity (DLTs) | within 4 weeks after infusion; 12, 24, 36 and 52 weeks after infusion
  To characterize the safety of anti-CD19 CAR NK Cells for moderate to severe refractory SLE
Incidence of Treatment Emergent Adverse Events (TEAEs) | within 4 weeks after infusion; 12, 24, 36 and 52 weeks after infusion
  To characterize the safety of anti-CD19 CAR NK Cells for moderate to severe refractory SLE

SECONDARY OUTCOMES:
SRI-4 response rate of subjects | 12, 24,36, and 52 weeks after infusion
  To characterize the efficacy of anti-CD19 CAR NK Cells for moderate to severe refractory SLE
LLDAS rate of subjects | 12, 24,36, and 52 weeks after infusion
  To characterize the efficacy of anti-CD19 CAR NK Cells for moderate to severe refractory SLE
DORIS remission rate of subjects | 12, 24,36, and 52 weeks after infusion
  To characterize the efficacy of anti-CD19 CAR NK Cells for moderate to severe refractory SLE

CONTACTS AND LOCATIONS:
Overall Officials: Dongbao Zhao, Doctor, Principal Investigator — ChanghaiHospital
Locations (1):
- Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gao J, Li M, Sun M, Yu Y, Kong R, Xu X, Liu S, Chen Q, Li X, Wu Y, Xu E, Yang J, Zhao D. Efficacy and safety of allogeneic CD19 CAR NK-cell therapy in systemic lupus erythematosus: a case series in China. Lancet. 2026 Dec 20;406(10522):2968-2979. doi: 10.1016/S0140-6736(25)01671-X. Epub 2025 Nov 12. PMID 41240964